CLINICAL TRIAL: NCT06608628
Title: The Effect of Patient Safety Escape Room on Nursing Students' Knowledge Level and Team Collaboration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Aysegul Yilmaz, Graduate Student, Karadeniz Technical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: KaradenızTekUnı
Record Dates: First submitted 2024-01-26; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Patient Safety
Keywords: Knowledge; Safety; Patient; Nursing Students; Collaboration; Gamification
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental and control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patient safety will play the escape room game.
  Interventions: Other: Experimental Group
- Control Group (Active Comparator): The control group will receive traditional training.
  .
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — The experimental group students will play a patient safety escape room game. Control group students will be given traditional education. The knowledge level and team cooperation of the two groups will be compared.
  Other Names: Control Group

SUMMARY:
The concept of patient safety first emerged more than two decades ago in research by practitioners applying different approaches to improve care in the areas they work in. The main goal in patient safety is to prevent mistakes while providing service, to protect patients from possible harm and to minimize the possibility of making mistakes. For this reason, patient safety is one of the indispensable parts of nursing education. The planned research will be carried out in order to increase the patient safety escape room design and the current knowledge level of student nurses and team cooperation on this subject. The research will be carried out with the first year students of the Faculty of Health Sciences, Nursing Department of a state university, in an experimental design with pre-test and post-test. The data of the research will be collected with the "General Information Questionnaire", "Patient Safety Knowledge Test", "Collaboration Scale" and "Gamy Experience for Gamification Scale". It is planned to carry out the study with 60 students. Control Group=30, Experiment Group=30. After the subject of patient safety is explained in the Nursing Fundamentals course, the students who agree to participate in the study will be randomly divided into experimental and control groups.

Patient safety practices will be explained to the control and experimental group students with the demonstration method in the laboratory environment after the lesson. Experimental group students will be taken to patient safety escape rooms prepared by the researcher. Students will be taken to escape rooms in groups of 5 and will be expected to perform the targeted tasks. After the lab and escape room activity, students will fill in the knowledge test and scales again. Since there is a limited number of studies in the literature on the knowledge levels of nursing students on patient safety and team collaboration, and there is no study in which escape room design is used in the field of nursing in Turkey, the research is important in terms of filling this gap in the literature.

DETAILED DESCRIPTION:
Nowadays, gamification not only improves knowledge levels positively, but also It is known that it is motivating and effective and increases the competitiveness of individuals. Moreover In gamification, it interrupts socialization, allows them to make mistakes, and provides immediate feedback. They provide advice and increase their technology. Use of games in nursing. It dates back to the 1980s. The use of gamification in education, optimization of in-class radiation, active problem-based learning and critical thinking characteristics in the growth in the learning process is developing. One of the games that has become popular in recent years is the escape room. escape room Games enable students to learn by experiencing and doing, based on problems. Also, your work. It increases their collaborative learning, motivation and knowledge level. Although escape room instructional design has been used in the international literature, there is no example used in Turkey. has not been found.

Therefore, the learning objective is based on the patient safety of student Sponsors through escape room instructional design. It combines levels of knowledge and business units of the team. Escape from Commercialism in Turkey There is no research involving room design, there is only systematic research on the subject. components and escape room game designs abroad, Reasons such as not including content are increasing the number of planned parts. also sick It has successes that evaluate the knowledge of its students regarding security. team collaboration. There are very few studies evaluating studies on official subjects. In the research literature. It will also be important to fill these sections.This research was conducted with Karadeniz Technical University Faculty of Health Sciences Nursing first year students will be done. The planned research will help student nurses learn about patient safety escape room game design. It will be carried out in order to increase the current knowledge levels and team cooperation on the subject. Escape Room permanent learning methods are used in its design. learning will be provided and students will have the opportunity to put the theoretical knowledge they have learned into practice. They will find it.

"General Information Survey", "Patient Safety Knowledge Test", "Workplace Information Test" were used as data collection tools in the research. Unity Scale" and "Gamelike Experience for Gamification Scale" will be used. Students After learning about patient safety within the scope of Nursing Fundamentals I course, participants were included in the study. Students who meet the admission criteria will be divided into two groups. Experimental group students escape from patient safety will be taken to their rooms. Control group students will continue traditional education. Before escape room and post-pre and post tests will be applied. After the room game, only the experimental group students were given "Gamelike Experience for Gamification scale" will be applied. In this study, students' patient safety knowledge scores, team cooperation. It is planned to increase their levels and determine their gaming experiences.

ELIGIBILITY:
Inclusion Criteria:

* Being a first year nursing student,
* Participating in a theoretical course on Patient Safety,
* Taking the Nursing Fundamentals-I course for the first time,
* Volunteering to participate in the research

Exclusion Criteria:

* Not attending the theoretical lecture on Patient Safety
* Nursing Fundamentals course have had it before
* Having transitioned to nursing through vertical transfer from other health departments,
* High school in a health-related field, Having an associate degree or bachelor's degree.
* Incomplete completion or failure to complete the pre-test or post-test,
* The student's wanting to withdraw from the research at some stage.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
HYPOTHESIS 1 | Two weeks
  Patient safety escape room has an impact on the knowledge level of nursing students.patient safety knowledge test.
HYPOTHESIS 2 | Two weeks
  Patient safety escape room has impact on the team cooperation level of nursing students.Scale of cooperation.
Research Question | Two weeks
  What are nursing students' patient safety escape room game experience scores?

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül Yılmaz,, Study Director — executive
Locations (1):
- Karadeniz Technical University, Trabzon, Kalkınma, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yilmaz A, Bayram SB. The effect of patient safety escape rooms on nursing students' knowledge level and team cooperation. Nurse Educ Pract. 2025 Aug;87:104507. doi: 10.1016/j.nepr.2025.104507. Epub 2025 Aug 13. PMID 40818273